CLINICAL TRIAL: NCT02018913
Title: Blood-brain Barrier Leakage in Dementia. A Dynamic Contrast-enhanced MRI Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Alzheimer Foundation (Other)
Responsible Party: Principal Investigator, F.R.J.Verhey, Professor of neuropsychiatry and old age psychiatry, Maastricht University Medical Center
Other Study IDs: NL46089.068.13
Record Dates: First submitted 2013-12-11; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease; Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Alzheimer's disease (AD) and vascular dementia (VaD) are the most common forms of dementia. Yet, the cause of these diseases is still unknown. A potentially important initiating factor is a disrupted blood-brain barrier. This can initiate cerebral microangiopathy, which has frequently been associated with VaD. Nevertheless, also in most AD patients a substantial increase of vascular damage has been observed. The present study investigates the correlation between blood-brain-barrier breakdown and cognitive decline in AD and VaD. An innovative dynamic contrast-enhanced MRI scan that has recently been developed and tested at our institute, will be used to measure blood-brain barrier permeability.

Objective: We will investigate the relationship between this permeability measure and (i) cognitive performance and (ii) the status of MRI visible cerebrovascular pathology (i.e. white matter hyperintensities, lacunar infarctions, microbleeds) in the most common forms of dementia.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Informed consent before participation in the study
* Age of 55 and older
* Diagnosed with AD, VaD, mixed AD and VaD, mild cognitive impairment, vascular cognitive impairment and subjective cognitive impairment
* MMSE ≥ 20 and patients are mentally competent (in general, individuals with an MMSE ≥18 are considered mentally competent)

Healthy participants:

* Informed consent before participation in the study
* Age of 55 and older
* No Diagnosis of dementia, prodromal dementia, or mild cognitive impairment.
* MMSE ≥ 26
* No substantial memory complaints (according to participant)
* Average age, gender and education is similar to the patient groups.

Exclusion Criteria:

* Contraindications for scanning (e.g. brain surgery, cardiac pacemaker, metal implants, claustrophobia, large body tattoos)
* Contraindications for contrast agent Gadovist (renal failure) as determined by the estimated Glomular Filtration Rate eGFR < 30 mL/min; or known allergy to Gadovist. If participants have a low renal function as determined by <30 GFR <60, the PI will contact a radiologist (Paul Hofman). The radiologist will decide if this patient should be excluded.
* Major vascular disorders (e.g. stroke, heart disease)
* Psychiatric or neurological disorders: Major depression (< 12 months); history of schizophrenia; bipolar disorder; psychotic disorder NOS or treatment for a psychotic disorder (< 12 mnd); cognitive impairment due to alcohol abuse; epilepsy; Parkinson's disease; MS; brain surgery; brain trauma; electroshock therapy; kidney dialysis; Meniere's disease; and brain infections.
* Structural abnormalities of the brain
* Cognitive impairment due to alcohol/drug abuse or abuse of other substances.
* Absence of reliable informant (for patient groups)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To obtain variation in macrovascular pathology and cognitive outcome measures, patients with AD, VaD, mixed AD and VaD, mild cognitive impairment (due to AD), vascular cognitive impairment and subjective cognitive impairment will be included. The total number of patients is 120, approximately 20 patients per disorder category as mentioned above. The patients will be recruited from the memory clinic of the Maastricht University Medical Center. Also a group of 20 age-matched healthy controls will be included. The total number of participants is thus 140.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Blood brain barrier permeability as measured by T1-weighted dynamic contrast MRI | Up to 4 years: April 2014-April 2018